CLINICAL TRIAL: NCT04086732
Title: Assessment of Generalized Alterations in Nociceptive Processing Among Patients Presenting With Temporo-mandibular Disorders
Brief Title: Assessment of Nociceptive Processing Among Patients With Temporo-mandibular Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HFS Mandibular
Record Dates: First submitted 2019-08-22; First posted 2019-09-12 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Temporomandibular Disorder
Keywords: central sensitization; high-frequency stimulation
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Temporomandibular disorder (Experimental)
  Interventions: Procedure: High-frequency electrical stimulation
- Healthy control (Experimental)
  Interventions: Procedure: High-frequency electrical stimulation

INTERVENTIONS:
Procedure: High-frequency electrical stimulation — High-frequency stimulation will be applied on the volar forearm (6-10 cm distal to the cubital fossa). To avoid any confounding effect of handedness, the arm onto which HFS will be applied twice (dominant vs nondominant) will be counterbalanced across participants. HFS will consist of 12 trains of 42 Hz electrical pulses lasting 1 s each. The time interval between each train will be 10 s. The intensity of stimulation will be milliampere. Electrical pulses will be delivered to the skin using a specifically-designed electrode designed: the cathode consists of 16 blunt stainless-steel pins with a diameter of 0.2 mm protruding 1 mm from the base. The 16 pins are placed in a circle with a diameter of 10 mm. The anode consists of a surrounding stainless-steel ring having an inner diameter of 22 mm and an outer diameter of 40 mm. This procedure induces secondary pinprick hyperalgesia (an increase in pinprick sensitivity in a large area of the skin).

SUMMARY:
This case control study will investigate the physiological effect of nociceptive input in individuals with temporomandibular disorders. To do so, the investigators will compare the development of secondary hyperalgesia following high frequency electrical stimulation (HFS) of skin nociceptors in the forearms for up to 48 hours in individuals with chronic TMD (as a main complain) and in healthy controls. Furthermore, the investigators will evaluate the association between the response to HFS and various factors, such as demographic, psychosocial and pain-related clinical factors.

DETAILED DESCRIPTION:
This control study is designed to compare the development of secondary hyperalgesia following high frequency electrical stimulation (HFS) of skin nociceptors in the forearms in individuals with chronic TMD (as a main complain) and in healthy controls.

During the first part of the experiment (time1, day 1), all potential participants will fill a basic demographic questionnaire concerning their age, weight, height, and current medications (appendix 2). Participants with TMD will be diagnosed according to the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD). The DC/TMD includes the following questionnaires: the Graded Chronic Pain Scale, the Jaw Functional Limitation scale, the Generalized Anxiety Disorder-7, the Patient Health Questionnaire-9 and -15 and the Oral Behaviors Checklist. In addition, participants will be asked to fill the Central sensitization inventory questionnaire, as well as the symptom Severity Scale. Lastly, the investigators will evaluate the distribution of pain by asking participants to draw the pain that they felt during the past 7 days on a digital tablet. This will allow us to determine the total area of pain of each participant, as well as the Widespread Pain Index. Subjects will also be asked to provide a rating of their average pain for the last 24h

The psychophysical evaluation will be conducted later on the same day (day1). Subjects will be asked to provide a rating of their average pain at present time (time 2). Then, participants will be familiarized with the different procedures involved in the experiment.

Pressure pain thresholds will be assessed on the temporalis muscle, the trapezius muscle, and tibialis anterior (time 3).

The intensity of pain resulting from pinprick stimulation and allodynia in the area surrounding the electrode ("test area") will be assessed, as well as on the homologous site of the contralateral control arm before HFS (time 4).

Then HFS will be applied (time 5) on the left or right volar forearm (10 cm distal to the cubital fossa). HFS will consist in trains of transcutaneous electrical stimuli consisting of 42 Hz trains (pulse width: 2 ms) lasting 1 s each. The trains will be repeated 12 times. Each train will be separated by several 10 seconds of rest. The intensity of each stimulus will be set to 5 milliampere.

The of pain resulting from pinprick stimulation and allodynia in the area surrounding the electrode ("test area") will be assessed 30 min after HFS (in a counterbalanced order) on the homologous site of the contralateral control arm (time 6).

The extent of secondary hyperalgesia will be assessed approximately 45 min following HFS (time 7).

Then, they will be asked assess the presence of secondary hyperalgesia in the test-site 24 (time 8, day 2) and 48 hours (time 9, day 3) following HFS with with calibrated neurological examination pins (Neuropen, Owen-Mumford Ltd, Oxford, UK).

6 months after their initial assessment (time 10, day 180), if they gave their consent for long-term follow-up, patients will be asked to fill the following questionnaires again

ELIGIBILITY:
Inclusion Criteria for healthy controls:

* Females aged between 18 and 50 years.
* BMI between 17 and 30.
* Ability to provide written informed consent.

Exclusion Criteria for healthy controls:

* Evidence of psychiatric/inflammatory/neurological or metabolic comorbidities on direct questioning as this study is meant to focus on musculoskeletal disorders.
* Evidence of skin alteration on the volar forearms that may interfere with HFS.
* Any substance abuse, or the use of antidepressant or neuroleptic medication as these may interfere with the psychophysical examination.
* Any painful musculoskeletal disorder.
* Lack of dental check-ups during the last 12 months.

Inclusion Criteria for the TMD group:

* Females aged between 18 and 50 years.
* BMI between 17 and 30.
* Ability to provide written informed consent.
* Chronic TMD (for at least 3 months) as a main complain (according to the DC/TMD), with an average of at least 3/10 on a pain numerical rating scale during the past month in the orofacial region.

Exclusion Criteria for the TMD group:

* Evidence of psychiatric/inflammatory/neurological or metabolic comorbidities on direct questioning as this study is meant to focus on musculoskeletal disorders.
* Evidence of skin alteration on the volar forearms that may interfere with HFS.
* Any substance abuse, or the use of antidepressant or neuroleptic medication as these may interfere with the psychophysical examination.
* Lack of dental check-ups during the last 12 months

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
The extent of secondary hyperalgesia on the forearm in the proximo-distal direction 45 minutes after HFS | After HFS and the assessment of pain resulting from pinprick stimulation and allodynia (time 7). This outcome is taken at day 1 at time 7.
  The area of secondary hyperalgesia (cm square) will be assessed with a calibrated 128 millinewton pinprick probe. Pokes of 1-second duration will be provided at a frequency of 0.5 Hz, starting well outside and approaching the stimulation site with steps of 0,5 cm from 4 different directions towards the application site. Participants will be asked to keep their eyes closed during the entire mapping procedure

SECONDARY OUTCOMES:
Age | During the initial evaluation (time 1). This outcome is taken at day 1 at time 1.
  Self-declared age of the subject
Weight | At baseline (time 1). This outcome is taken at day 1 at time 1.
  Self-declared weight of the subject
Height | At baseline (time 1). This outcome is taken at day 1 at time 1.
  Self-declared height of the subject
The TMD diagnosis according to the diagnostic criteria for temporomandibular disorders (DC/TMD) | At baseline (time 1). This outcome is taken at day 1 at time 1.
  TMD subgroup based on the DC/TMD: Myalgia, Arthralgia, Headache attributed to TMD, degenerative joint disease, disc displacement with reduction, disc displacement with reduction with intermittent locking, disc displacement with reduction with limited opening, disc displacement with reduction without limited opening, or subluxation.
Graded chronic pain scale | At baseline (time 1) and 6 months after the initial assessment (time 10). This outcome is taken at day 1 at time 1 and day 180 at time 10.
  questionnaire assessing TMD-related pain intensity and disability: The score will range from grade 0 (no TMD pain in prior 6 months) to grade IV (High disability, severly limiting)
Jaw functional limitation scale | At baseline (time 1) and 6 months after the initial assessment (time 10). This outcome is taken at day 1 at time 1 and day 180 at time 10.
  Questionnaire assessing limitations across mastication, jaw mobility, and verbal and emotional expression often accompanying TMD. The score will range from 0 (law functional limitation) to 10 (high functional limitation)
Generalized anxiety disorder-7 | At baseline (time 1) and 6 months after the initial assessment (time 10). This outcome is taken at day 1 at time 1 and day 180 at time 10.
  Questionnaire assessing anxiety. The score will range from 0 (no anxiety) to 27 (severe anxiety)
Patient health questionnaire-9 | At baseline (time 1) and 6 months after the initial assessment (time 10). This outcome is taken at day 1 at time 1 and day 180 at time 10.
  Questionnaire assessing depression symptoms. The score will range from 1 (minimal depression) to 27 (severe depression)
Patient health questionnaire-15 | At baseline (time 1) and 6 months after the initial assessment (time 10). This outcome is taken at day 1 at time 1 and day 180 at time 10.
  Questionnaire assessing overall physical symptoms commonly associated with TMD. The score will range from 0 (minimal physical symptoms) to 30 (high physical symptoms)
Oral Behaviors Checklist | At baseline (time 1) and 6 months after the initial assessment (time 10). This outcome is taken at day 1 at time 1 and day 180 at time 10.
  Questionnaire assesses the frequency of oral parafunctional behaviors. The score will range from 0 (no oral parafunctional behaviors) to 84 (high oral parafunctional behavior frequency)
Central sensitization inventory | At baseline (time 1) and 6 months after the initial assessment (time 10). This outcome is taken at day 1 at time 1 and day 180 at time 10.
  Questionnaire assessing symptoms and comorbidities that are presumed to be associated with central sensitization. The score will range from 0 (no symptoms and comorbidities presumed to be associated with central sensitization) to 100 (extreme symptoms and comorbidities presumed to be associated with central sensitization).
Symptom severity scale | At baseline (time 1) and 6 months after the initial assessment (time 10). This outcome is taken at day 1 at time 1 and day 180 at time 10.
  Questionnaire assessing the severity of symptoms associated with fibromyalgia, a condition frequently associated with TMD. The score will range from 0 (low severity) to 12 (high severity).
The distribution of pain | At baseline (time 1) and 6 months after the initial assessment (time 10). This outcome is taken at day 1 at time 1 and day 180 at time 10.
  Pain felt during the past 7 days drawn on a digital table
The Widespread pain index | At baseline (time 1) and 6 months after the initial assessment (time 10). This outcome is taken at day 1 at time 1 and day 180 at time 10.
  Questionnaire assessing the extent of bodily pain. The score will range from 1 (no painful body region) to 19 (19 painful body regions)
Average pain during the last 24h before HFS | During the initial evaluation (time 1). This outcome is taken at day 1 at time 1.
  Pain during the last 24h on a numerical rating scale. The score will range from 0 (no pain) to 100 (worst imaginable pain)
Average pain at present time before HFS: score | During the initial evaluation (time 2). This outcome is taken at day 1 at time 2.
  Current pain on a numerical rating. The score will range from 0 (no pain) to 100 (worst imaginable pain)
Pressure pain thresholds on the temporalis muscle, trapezius muscle and tibialis anterior | During the initial evaluation (time 3)]. This outcome is taken at day 1 at time 3.
  Pressure pain will be assessed 3 times on each muscle, with a 30-second interstimulus interval, and the arithmetic mean of the 3 repeated measures will be used for analysis
Baseline pain resulting from pinprick stimulation in the area surrounding the electrode ("test area") and on the homologous site of the contralateral control arm | Just before HFS (time 4)]. This outcome is taken at day 1 at time 4.
  Participants will rate the pain induced by pin-prick stimulation in the area surrounding the electrode on a numerical rating scale ranging from 0 (no perception) to 100 (maximal pain), with 50 representing the transition from nonpainful to painful domains of sensation
Allodynia in the area surrounding the electrode ("test area") and on the homologous site of the contralateral control arm | Just before HFS (time 4) and after HFS (time 6). This outcome is taken at day 1 at time 4 and time 6.
  The investigators will assess allodynia with a Cotton wisp exerting a force of 3 millinewton, a cotton wool tip fixed to an elastic strip exerting a force of 100 millinewton when slightly bent, and a standardized brush exerting a force of 200-400 millinewton
The long term persistence of secondary hyperalgesia after HFS | 24 hours (time 8) and 48 hours after HFS (time 9). This outcome is taken at day 2 at time 8, and at day 3 at time 9.
  Participants will assess the persistence of secondary hyperalgesia with calibrated neurological examination pins (Neuropen, Owen-Mumford Ltd, Oxford, UK). The score will range from 0 (no hyperalgesia) to 1 (hyperalgesia is present)
The intensity of pain resulting from pinprick stimulation 30 min after HFS | Time Frame: At baseline (time 6). This outcome is taken at day 1 at time 6.
  Participants will rate the pain induced by pin-prick stimulation in the area surrounding the electrode on a numerical rating scale ranging from 0 (no perception) to 100 (maximal pain), with 50 representing the transition from nonpainful to painful domains of sensation

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires St-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No